CLINICAL TRIAL: NCT06153511
Title: Clinical Investigation With a Robotic Assistant for Spinal Surgery in Patients Requiring a Transpedicular Fixation
Brief Title: Clinical Study With a Robotic Assistant in Patients Requiring a Spinal Transpedicular Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyber Surgery S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROTCL-CYB-01-PIC
Record Dates: First submitted 2023-11-16; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: SPINAL Fracture; Vertebral Fractures; Spinal Stenosis; Kyphosis; Lumbar Spinal Stenosis; Thoracolumbar Kyphosis
Keywords: Robot assisted spinal fusion
MeSH Terms: conditions — Spinal Fractures; Spinal Stenosis; Kyphosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with spinal condition who requires a transpedicular fixation intervention. (Experimental): Patient with spinal condition (vertebral fractures, spinal stenosis, kyphosis, among others) who requires a intervention for spinal fusion with pedicle screws.
  Interventions: Procedure: Robot assisted spinal transpedicular fixation

INTERVENTIONS:
Procedure: Robot assisted spinal transpedicular fixation — Surgical technique which joins two or more vetebrae with screws and rods to prevent any relative movement between them. It is a major surgery that usually lasts several hours and in which the patient is subjected to general anesthesia. The screws to be placed go through a narrow area of the vertebra known as the pedicle. Each patient will undergo a singular intervention.
  Other Names: Robotic assisted pedicle screw insertion

SUMMARY:
This multicenter, non-comparative clinical trial, led by two principal investigators in Spain, aims to evaluate the safety and performance of a robotic assistant, based on a electromechanical tracking system, in patients requiring transpedicular screw fixation. The study, conducted in two different hospital centers, involves patients with vertebral fractures, spinal stenosis, kyphosis, and other related conditions. The primary objective is to determine screw accuracy by assessing the degree of screw invasion into the pedicle using the Gertzbein-Robbins scale, with a target of achieving 96% acceptable screw placement. Trained radiologists will evaluate the screw invasion into the pedicle. The study is scheduled to span 12 months and each intervention includes a 1-month follow-up. Throughout this time frame, patients will undergo regular assessments, and outcomes will be closely monitored.

DETAILED DESCRIPTION:
Multicenter non-comparative clinical trial.

This interventional study aims to assess the safety and performance of a robotic assistant, based on a electromechanical tracking system, in patients requiring transpedicular screw fixation.The primary focus is on overcoming the limitations of traditional minimally invasive surgeries and enhancing the accuracy of pedicle screw placement, especially within the complex pedicle region adjacent to the spinal canal.

The study design is a prospective interventional trial conducted in two hospital centers in Spain, with two principal investigators leading the investigation. Patients requiring transpedicular screw fixation will be recruited. The robotic assistant will be employed to facilitate transpedicular screw fixation. The system aims to improve accuracy and safety in screw placement, in comparison with conventional techniques used.

Patients will include individuals with spinal fractures, spinal stenosis, kyphosis, and other conditions requiring transpedicular screw fixation. Two principal investigators in Spain will lead the recruitment process.

The study aims to answer several key questions:

* Determine Screw Accuracy: Assess the degree of screw invasion into the pedicle using the Gertzbein-Robbins scale, with a target of achieving 96% acceptable screw placement.
* Evaluate Planning vs. Final Screw Placement: Determine the accuracy of screw placement by comparing planned positions with the actual final positions.
* System Performance: Assess the overall performance of the robotic system during the surgical procedure.
* Reoperation and Postoperative Time: Determine the need for reoperation and evaluate postoperative recovery time.
* Adverse Events: Detect and document any adverse events occurring during the surgical process.

Trained radiologists will play a crucial role in evaluating the accuracy of screw placement, focusing on the degree of invasion into the pedicle using the Gertzbein-Robbins scale. The study is set to span a duration of 12 months,during which patients will undergo regular assessments, and outcomes will be closely monitored. The inclusion of the electromechanical tracking system in the robotic assistant adds a technological dimension to the investigation, contributing to advancements in the field of minimally invasive spinal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for spinal fusion Surgery requiring pedicle screw insertion.
* Open or minimally invasive (MIS) technique.
* Spinal regions: lumbar, thoracic and/or sacral (one patient may cover several regions).
* Signed informed consent.

Exclusion Criteria:

* Paediatric patient (< 18 years)
* Pedicular Surgery history with screw insertion in the vertebra to be operated.
* Any contraindication for the pedicular screw placement.
* Severe scoliosis.
* Severe osteoporosis.
* Infection or neoplasia.
* Obesity.
* Pregnancy and lactancy.
* Any other disease or disorder that, in the opinión of the neurosurgeron, may put the patient at risk or may influence the results of the study.
* Simultaneous participation in other clinical studies.
* For whatever reason, the Clinical protocol cannot be followed.
* The patient is unable, or unwilling, to sign the informed consent.
* Patients in emergency situation who are not legally able to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Grade of screw invasion into the pedicle based on Gertzbein-Robbins scale (A-E grade) | 1 month follow-up
  Grade A: Screw position within the pedicle. Grade B: Cortical breakage ≤2mm. Grade C: Cortical breakage ≤4mm. Grade D: Cortical breakage ≤6mm. Grade E: Cortical breakage >6mm.

SECONDARY OUTCOMES:
Patient characteristics - Demographic dates - Sex (Male/Female) | 3 months
Patient characteristics - Demographic dates - Age (years) | 3 months
Patient characteristics - Demographic dates - Weight (kg) | 3 months
Patient characteristics - Demographic dates - Height (cm) | 3 months
Patient characteristics - BMI | 3 months
  W [kg]/H [m2]
Patient characteristics - Spinal Region (Thoracic/Lumbar/Sacral) | 3 months
Patient characteristics - Vertebrae for study (T1...T12/L1...L5/S1-S2) | 3 months
Patient characteristics - Comobidities | 3 months
  Charlson Index (1-6 pts)
Patient characteristics - Number of screws to be placed | 3 months
Implant characteristics - Planned vertebrae | 3 months
Implant characteristics - Laterality (L/R) | 3 months
Implant characteristics - Screw orientation in sagittal plane (Cranial/Caudal/Neutral) | 3 months
Implant characteristics - Screw orientation in axial plane (Medial/Lateral/Neutral) | 3 months
Implant characteristics - Screw dimensions - Screw diameter (mm) | 3 months
Implant characteristics - Screw dimensions - Screw length (mm) | 3 months
Clinical Intervention - Surgical technique (open/MIS) | 3 months
Clinical Intervention - ASA Anaesthesia (I-IV) | 3 months
Clinical Intervention - Radiation emission - Time (sec.) | 3 months
Clinical Intervention - Radiation emission - Dosage (mGy) | 3 months
Clinical Intervention - Blood loss - Intraoperatice blood loss (ml) | 3 months
Clinical Intervention - Blood loss - Number of gauzes used | 3 months
Clinical Intervention - Blood loss - Postoperative drainage (ml) | 3 months
Clinical Intervention - Blood loss - Duration of surgery - Total (min.) | 3 months
Clinical Intervention - Blood loss - Duration of surgery per stages - Power on and disposition (min.) | 3 months
Clinical Intervention - Blood loss - Duration of surgery per stages - Planification (min.) | 3 months
Clinical Intervention - Blood loss - Duration of surgery per stages - Image registration (min.) | 3 months
Clinical Intervention - Blood loss - Duration of surgery per stages - Positioning (min.) | 3 months
Clinical Intervention - Blood loss - Duration of surgery per stages - Surgery (min.) | 3 months
Clinical Intervention - Blood loss - Duration of surgery per stages - Removal and power off (min.) | 3 months
Clinical Intervention - Blood loss - Postoperative stay (days) | 1 month follow-up
System performance - Number of image registration | 1 month follow-up
System performance - Number of screws not inserted using the robotic assistant | 1 month follow-up
System performance - Number of colisioned screws | 1 month follow-up
System performance - Number of not reachable screws | 1 month follow-up
System performance - Fiducial Registration Error, FRE (mm) | 3 months
System performance - Screw position deviation - Spatial deviation in XY plane (mm) | 1 month follow-up
System performance - Screw position deviation - Spatial deviation in XZ plane (mm) | 1 month follow-up
System performance - Screw position deviation - Spatial deviation in YZ plane (mm) | 1 month follow-up
System performance - Screw position deviation - Angular deviation in XY plane (deg.) | 1 month follow-up
System performance - Screw position deviation - Angular deviation in XZ plane (deg.) | 1 month follow-up
System performance - Screw position deviation - Angular deviation in YZ plane (deg.) | 1 month follow-up
Adverse Events, AE | 1 month follow-up
Severe Adverse Events, SAE | 1 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nicolás M. Samprón Lebed, Neurosurgeon, Principal Investigator — Hospital Donostia; Iñigo C. Pomposo Gastelu, Neurosurgeon, Principal Investigator — Hospital de Cruces
Locations (1):
- Cyber Surgery, Donostia / San Sebastian, Gipuzkoa, Spain

IPD SHARING:
Plan to Share IPD: No